CLINICAL TRIAL: NCT03785678
Title: A Phase III, Prospective, Double-blind, Randomized, Placebo-controlled Trial of Thrombolysis in Imaging-eligible, Late-window Patients to Assess the Efficacy and Safety of Tenecteplase (TIMELESS)
Brief Title: Tenecteplase in Stroke Patients Between 4.5 and 24 Hours
Acronym: TIMELESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ML40787
Record Dates: First submitted 2018-12-19; First posted 2018-12-24 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: THROMBOLYSIS
MeSH Terms: interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tenecteplase (Experimental): Patients in this arm will receive Tenecteplase (0.25 mg/kg, maximum 25 mg) administered as a single bolus injection over 5 seconds.
  Interventions: Biological: Tenecteplase
- Placebo (Placebo Comparator): Patients in this arm will receive placebo administered as a single bolus injection over 5 seconds.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tenecteplase — The investigational medicinal product (IMP) for this study is tenecteplase. The recommended total dose for this study is weight-based with 0.25 mg of tenecteplase per kg, not exceeding a maximum dose of 25 mg. A single bolus dose should be administered over 5 seconds based on patient weight.
  Arms: Tenecteplase
Other: Placebo — Placebo is being used as the comparator since a thrombolytic is only FDA-approved in the United States for use out to 3 hours, and the standard of care guidelines support use out to 4.5 hours.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of tenecteplase compared with placebo in participants with acute ischemic stroke (AIS).

All participants will receive standard-of-care therapy according to AmericanHeart Association/American Stroke Association clinical guidelines (2018). To determine eligibility for randomization, all participants will undergo multimodal CT or MRI at baseline. Only participants with a vessel occlusion (ICA or MCA M1/M2) and penumbral tissue will be randomized. The primary analysis is to compare the efficacy of tenecteplase versus placebo in all participants at Day 90.

ELIGIBILITY:
Inclusion Criteria:

* Patient/legally authorized representative has signed the Informed Consent Form
* Age >= 18 years
* AIS symptom onset within 4.5 to 24 hours Signs and symptoms consistent with the diagnosis of an acute anterior circulation ischemic stroke involving occlusion of the ICA, M1, or M2 vessels
* Functionally independent (mRS 0-2) prior to stroke onset
* Baseline NIHSS >=5 and that remains >=5 immediately prior to randomization
* Neuroimaging: ICA or M1, M2 occlusion (carotid occlusions can be cervical or intracranial, with or without tandem MCA lesions) by magnetic resonance angiography (MRA) or computed tomography angiography (CTA) AND target mismatch profile on CT perfusion or MR perfusion (ischemic core volume <70 mL, mismatch ratio is >=1.8 and mismatch volume is >= 15 mL)
* The mismatch volume is determined by FDA-approved imaging software in real time based on the difference between the ischemic core lesion volume and the Tmax>6s lesion volume. If both a CT perfusion and a multimodal MRI scan are performed prior to enrollment, the later of the 2 scans is assessed to determine eligibility. Only an intracranial MRA is required for patients screened with MRA; cervical MRA is not required. Cervical and intracranial CTA are typically obtained simultaneously in patients screened with CTA, but only the intracranial CTA is required for enrollment.

Alternative neuroimaging:

* If CTA (or MRA) is technically inadequate: Tmax>6s perfusion deficit consistent with an ICA or M1, M2 occlusion AND target mismatch profile (ischemic core volume <70 mL, mismatch ratio >= 1.8 and mismatch volume >= 15 mL as determined by RAPID software)
* If magnetic resonance perfusion (MRP) is technically inadequate: ICA or M1, M2 occlusion (carotid occlusions can be cervical or intracranial; with or without tandem MCA lesions) by MRA (or CTA, if MRA is technically inadequate and a CTA was performed within 60 minutes prior to the MRI) AND diffusion-weighted imaging (DWI) lesion volume <=25 mL for an M1 or ICA occlusion and =<15 mL for an M2 occlusion
* If CTP is technically inadequate: patient can be screened with MRI and randomized if neuroimaging criteria are met.
* Ability to comply with the study protocol, in the investigator's judgment

Exclusion Criteria:

General

* Current participation in another investigational drug or device study
* Active internal bleeding
* Known hypersensitivity or allergy to any ingredients of tenecteplase
* Known bleeding diathesis
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; recent oral anticoagulant therapy with INR >1.7
* Use of one of the new oral anticoagulants within the last 48 hours (dabigatran, rivaroxaban, apixaban, edoxaban)
* Pregnant
* Intracranial neoplasm (except small meningioma), arteriovenous malformation, or aneurysm
* Seizures at stroke onset if it precludes obtaining an accurate baseline NIHSS
* Severe, uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure > 110 mmHg)
* For participants with suspected coagulopathy, platelet count must be checked prior to randomization and participant is excluded if baseline platelet count <100,000/microL
* Baseline blood glucose >400 mg/dL (22.20 mmol/L)
* Baseline blood glucose <50 mg/dL needs to be normalized prior to randomization
* Clot retrieval attempted using a neurothrombectomy device prior to randomization
* Intracranial or intraspinal surgery or trauma within 2 months
* Treatment with a thrombolytic within the last 3 months prior to randomization
* Other serious, advanced, or terminal illness (investigator judgment) with life expectancy less than 6 months
* Pre-existing medical, neurological, or psychiatric disease that would confound the neurological or functional evaluations
* History of cerebrovascular accident in the last 90 days
* Presumed septic embolus; suspicion of bacterial endocarditis
* Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the patient if an endovascular procedure was to be performed

Imaging

* Unable to undergo a contrast brain perfusion scan with either MRI or CT
* Extensive early ischemic change (hypodensity) on non-contrast CT estimated to be >1/3 MCA territory, or significant hypodensity outside the Tmax>6s perfusion lesion that invalidates mismatch criteria (if patient is enrolled based on CT perfusion criteria)
* Significant mass effect
* Acute symptomatic arterial occlusions in more than one vascular territory confirmed on CTA/MRA (e.g., bilateral MCA occlusions, or an MCA and a basilar artery occlusion)
* Evidence of intracranial tumor (except small meningioma) acute intracranial hemorrhage, neoplasm, or arteriovenous malformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (97):
- United States (94):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Desert Medical Center, Mesa, Arizona
  - Kaiser Permanente - Anaheim (E. La Palma), Anaheim, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - John Muir Health, Concord Medical Center, Concord, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente - Fontana, Fontana, California
  - Adventist Health Glendale, Glendale, California
  - Kaiser Permanente South Bay Medical Center, Harbor City, California
  - UCSD Medical Center - La Jolla, La Jolla, California
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - University of Southern California Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Cedars-Sinai Marina Del Rey Hospital, Marina del Rey, California
  - Kaiser Permanente - Ontario, Ontario, California
  - Stanford University Medical Center, Palo Alto, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Group, Neurology, Sacramento, California
  - UCSD - Hillcrest; Hillcrest Medical Center, San Diego, California
  - CPMC - Van Ness Campus, San Francisco, California
  - CPMC - Davies Campus, San Francisco, California
  - Torrance Memorial Medical Center, Torrance, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida Health at Shands, Gainesville, Florida
  - Baptist Medical Center - Jacksonville, Jacksonville, Florida
  - Baptist Medical Center-South, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - St. Catherine Hospital, East Chicago, Indiana
  - St. Mary Medical Center, Hobart, Indiana
  - Community Hospital, Munster, Indiana
  - Uni of Kansas Medical Center, Kansas City, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Univ of Michigan Medical Ctr, Ann Arbor, Michigan
  - Henry Ford Macomb Hospital - Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Flint, Flint, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - ProMedica Monroe Regional Hospital, Monroe, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Fairview Southdale, Edina, Minnesota
  - U of Minnesota MedCtr Fairview, Minneapolis, Minnesota
  - Sanford Worthington Medical Center, Worthington, Minnesota
  - Washington University, St Louis, Missouri
  - JFK Neuroscience Institute, Edison, New Jersey
  - Atlantic Health System - Overlook Medical Center, Summit, New Jersey
  - Capital Health Regional Medical Center, Trenton, New Jersey
  - Buffalo General Medical Center, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Mission Hospitals Inc, Asheville, North Carolina
  - Guilford Neurologic Research, Greensboro, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Riverside Methodist Hospital; Cancer Services, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Ascension St. John, Tulsa, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Health Portland, Portland, Oregon
  - Providence Saint Vincent's Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - UPMC East Hospital, Monroeville, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Uni of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UPMC Mercy, Pittsburgh, Pennsylvania
  - UPMC Passavant Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Sanford Neurology Clinic, Sioux Falls, South Dakota
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - Saint Thomas Rutherford Hospital, Murfreesboro, Tennessee
  - Saint Thomas Health, Nashville, Tennessee
  - Saint Thomas Midtown Hospital, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Dell Seton Medical center at the University of Texas, Austin, Texas
  - Seton Medical Center Austin, Austin, Texas
  - Valley Baptist Medical Center-Brownsville, Brownsville, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Valley Baptist Medical Center, Harlingen, Texas
  - University of Texas at Houston; Neurology, Houston, Texas
  - Ascension Seton Hays, Kyle, Texas
  - Ascension Seton Williamson, Round Rock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
- Canada (3):
  - Uni of Alberta, Edmonton, Alberta
  - Hamilton General Hospital; Pharmacy, Hamilton, Ontario
  - Montreal Neurological Inst; Clinical Research Unit, Montreal, Quebec

REFERENCES:
- [Derived] Albers GW, Jumaa M, Purdon B, Zaidi SF, Streib C, Shuaib A, Sangha N, Kim M, Froehler MT, Schwartz NE, Clark WM, Kircher CE, Yang M, Massaro L, Lu XY, Rippon GA, Broderick JP, Butcher K, Lansberg MG, Liebeskind DS, Nouh A, Schwamm LH, Campbell BCV; TIMELESS Investigators. Tenecteplase for Stroke at 4.5 to 24 Hours with Perfusion-Imaging Selection. N Engl J Med. 2024 Feb 22;390(8):701-711. doi: 10.1056/NEJMoa2310392. Epub 2024 Feb 8. PMID 38329148
- [Derived] Zachrison KS, Amati V, Schwamm LH, Yan Z, Nielsen V, Christie A, Reeves MJ, Sauser JP, Lomi A, Onnela JP. Influence of Hospital Characteristics on Hospital Transfer Destinations for Patients With Stroke. Circ Cardiovasc Qual Outcomes. 2022 May;15(5):e008269. doi: 10.1161/CIRCOUTCOMES.121.008269. Epub 2022 Apr 4. PMID 35369714
- [Derived] Albers GW, Campbell BC, Lansberg MG, Broderick J, Butcher K, Froehler MT, Schwamm LH, Nouh AM, Liebeskind DS, Toy F, Yang M, Massaro L, Schoeffler M, Purdon B. A Phase III, prospective, double-blind, randomized, placebo-controlled trial of thrombolysis in imaging-eligible, late-window patients to assess the efficacy and safety of tenecteplase (TIMELESS): Rationale and design. Int J Stroke. 2023 Feb;18(2):237-241. doi: 10.1177/17474930221088400. Epub 2022 Apr 1. PMID 35262424

RESULTS

PARTICIPANT FLOW:
Groups:
- Tenecteplase: Participants received Tenecteplase (0.25 mg/kg, maximum 25 mg) administered as a single bolus injection over 5 seconds, administered within 4.5 - 24 hours of the onset of internal carotid artery (ICA) or middle cerebral artery (MCA) stroke.
- Placebo: Participants received placebo administered as a single bolus injection over 5 seconds, administered within 4.5 - 24 hours of the onset of internal carotid artery (ICA) or middle cerebral artery (MCA) stroke.
Period: Overall Study
Arm/Group | Tenecteplase | Placebo
Started | 228 | 230
Completed | 175 | 181
Not Completed | 53 | 49
Not completed — Death | 44 | 42
Not completed — Lost to Follow-up | 4 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenecteplase | Placebo | Total
Number analyzed (Participants) | 228 | 230 | 458
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (13.5) | 71.3 (13.6) | 70.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 123 | 245
  Male | 106 | 107 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 22 | 39
  Not Hispanic or Latino | 201 | 197 | 398
  Unknown or Not Reported | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 11 | 9 | 20
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 31 | 32 | 63
  White | 169 | 170 | 339
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Ordinal Modified Rankin Scale (mRS) Score at Day 90
Description: The the modified Rankin score (mRS) is a 6-point scale commonly used to assess disability due to stroke, with higher values indicating worse outcomes.
  0 = No symptoms
  1. = No significant disability
  2. = Slight disability
  3. = Moderate disability
  4. = Moderately severe disability
  5. = Severe disability
  6. = Death
Time Frame: Day 90
Population: The ITT population consisted of all randomized participants who provided informed consent, with participants grouped according to their assigned treatment.
Measure: Number; unit: Count of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 226 | 229
Count of participants
  0 | 35 | 31
  1 | 38 | 30
  2 | 31 | 36
  3 | 34 | 41
  4 | 29 | 34
  5 | 15 | 13
  6 | 44 | 44

2. Secondary Outcome: Proportion of Patients With Functional Independence at Day 90
Description: Functional independence, was defined as an mRS of 0-2 (no symptoms to mild symptoms), at Day 90.
Time Frame: Day 90
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 226 | 229
Percentage of participants
  mRS ≤ 2 at Day 90 | 46.0 | 42.4
  mRS > 2 at Day 90 | 54.0 | 57.6

3. Secondary Outcome: Proportion of Patients With Recanalization at 24 Hours Post-randomization
Description: This endpoint measured complete or partial recanalization (restored blood flow) on CT angiography (CTA)/magnetic resonance angiography (MRA) post-randomization, defined as complete or partial recanalization on CT angiography (CTA)/magnetic resonance angiography (MRA).
Time Frame: Day 2
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 193 | 194
Percentage of participants
  Complete recanalization | 76.7 | 63.9
  None or partial recanalization | 23.3 | 36.1

4. Secondary Outcome: Proportion of Patients With Reperfusion at 24 Hours Post-randomization
Description: This endpoint was defined by the proportion of participants with reperfusion (the restoration of blood flow to an organ or tissue after having been blocked) at 24 hours post-randomization, defined as > 90% reduction in Tmax > 6s lesion volume.
Time Frame: Day 2
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 174 | 182
Percentage of participants
  > 90% reduction in Tmax > 6s lesion volume | 56.9 | 57.7
  ≤ 90% reduction | 43.1 | 42.3

5. Secondary Outcome: Proportion of Patients With Angiographic Reperfusion at Completion of Angiographic Procedure
Description: Angiographic reperfusion was evaluated using the modified Thrombolysis in Cerebral Infarction (TICI) Scale:
  0: No perfusion or anterograde flow beyond site of occlusion.
  1. Contrast passes the area of occlusion but fails to opacify the entire cerebral bed distal to the obstruction during angiographic run.
  2. Partial perfusion wherein the contrast passes the occlusion and opacifies the distal arterial bed but rate of entry or clearance from the bed is slower than non-involved territories 2A: < 50% of territory visualized 2B: ≥ 50% of territory is visualized 2C: Near complete perfusion except for slow flow in a few distal cortical vessels or presence of small distal cortical emboli
  3. Complete reperfusion with normal filling.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 175 | 178
Percentage of participants
  Achieving TICI 2b or TICI 3 | 89.1 | 85.4
  Achieving TICI < 2b | 10.9 | 14.6

6. Secondary Outcome: Median NIHSS Score at Day 90
Description: The National Institutes of Health Stroke Score (NIHSS) is a 15-item scale that measures neurological deficit in acute stroke patients. Each item is ranked using a 3-, 4-, or 5-point scale, including allowances for items that cannot be scored due to the patient's condition, with higher scores indicating more severe deficit. Total scores range from 0-42, with higher scores indicating more severe deficits.
Time Frame: Day 90
Population: as for outcome 1
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 79 | 89
Scores on a scale | 1.0 [0 to 31] | 1.0 [0 to 26]

7. Secondary Outcome: Proportion of Patients With a Barthel Index (BI) Score ≥ 95 at Day 90
Description: The Barthel Index (BI) is a 10-item ordinal scale used to measure performance in activities of daily living (ADL) and mobility. The BI scoring range is from 0-100, with lower scores representing greater dependency.
Time Frame: Day 90
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 81 | 89
Percentage of participants
  BI score ≥ 95 at Day 90 | 60.5 | 58.4
  BI score < 95 at Day 90 | 39.5 | 41.6

8. Secondary Outcome: Proportion of Patients With Good Recovery Based on the Glasgow Outcome Scale (GOS) at Day 90
Description: The Glasgow Outcome Scale (GOS) is a scale used to assess recovery of participants with brain damage. The scale has 5 categories:
  1. = Death
  2. = Persistent vegetative state
  3. = Severe disability
  4. = Moderate disability
  5. = Good recovery
  The GOS was re-scaled from observed data. For this measure, 1 = good recovery and 5 = death.
Time Frame: Day 90
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 126 | 133
Percentage of participants
  Good recovery GOS score (=1) | 36.5 | 30.8
  GOS score > 1 | 63.5 | 69.2

9. Secondary Outcome: Incidence of Symptomatic Intracranial Hemorrhage (sICH) Within 36 Hours
Time Frame: Within 36 hours (Day 2) of treatment
Population: The safety population consisted of all randomized participants who received tenecteplase or placebo, with participants grouped according to the treatment actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 218 | 214
Percentage of participants | 3.2 | 2.3

10. Secondary Outcome: Mortality Rate up to Day 30 and Day 90
Time Frame: Day 30 and Day 90
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 218 | 214
Percentage of participants
  Death within 30 days | 14.7 | 15.0
  Death within 90 days | 19.7 | 18.2

11. Secondary Outcome: Proportion of Patients With Parenchymal Hematoma Type 2 (PH2) at the 72-96 Hour Visit
Time Frame: Day 3
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 218 | 214
Percentage of participants | 3.7 | 2.8

ADVERSE EVENTS:
Time Frame: From treatment visit to Day 90 follow-up
Description: All-cause mortality was assessed for all participants.
  Serious Adverse Events and Other Adverse Events were assessed for the safety population, which consisted of all randomized participants who received tenecteplase or placebo, with participants grouped according to the treatment actually received.
Arm/Group | Tenecteplase | Placebo
All-Cause Mortality (participants affected / at risk) | 44/228 | 44/230
Serious Adverse Events (participants affected / at risk) | 91/218 | 102/214
Other Adverse Events (participants affected / at risk) | 145/218 | 136/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenecteplase (N=218) | Placebo (N=214)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 4 (4)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac arrest (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2)
Death (General disorders) | 2 (2) | 3 (3)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 4 (4) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 6 (6)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
NIH stroke scale abnormal (Investigations) | 0 (0) | 1 (1)
Neurological examination abnormal (Investigations) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 7 (7) | 2 (2)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery perforation (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 5 (5) | 7 (7)
Cerebral artery perforation (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral haemorrhage (Nervous system disorders) | 4 (4) | 3 (4)
Cerebral infarction (Nervous system disorders) | 2 (2) | 3 (4)
Cerebrovascular accident (Nervous system disorders) | 6 (7) | 7 (7)
Cerebrovascular disorder (Nervous system disorders) | 2 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 3 (3)
Haemorrhage intracranial (Nervous system disorders) | 4 (4) | 5 (5)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 5 (5) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 3 (3)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 1 (1) | 2 (2)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 2 (2)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Stroke in evolution (Nervous system disorders) | 7 (7) | 13 (13)
Subarachnoid haemorrhage (Nervous system disorders) | 6 (6) | 4 (4)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (2)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (8)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Arterial aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Therapy cessation (Surgical and medical procedures) | 1 (1) | 0 (0)
Air embolism (Vascular disorders) | 2 (2) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (3)
Distributive shock (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 8 (8) | 0 (0)
Labile blood pressure (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery haematoma (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenecteplase (N=218) | Placebo (N=214)
Anaemia (Blood and lymphatic system disorders) | 13 (13) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 12 (12) | 18 (19)
Constipation (Gastrointestinal disorders) | 13 (13) | 13 (13)
Dysphagia (Gastrointestinal disorders) | 13 (13) | 5 (5)
Pyrexia (General disorders) | 12 (12) | 15 (16)
Pneumonia (Infections and infestations) | 12 (12) | 6 (6)
Urinary tract infection (Infections and infestations) | 29 (31) | 20 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (19) | 27 (27)
Cerebral haemorrhage (Nervous system disorders) | 22 (22) | 13 (13)
Haemorrhage intracranial (Nervous system disorders) | 14 (14) | 10 (11)
Haemorrhagic transformation stroke (Nervous system disorders) | 28 (29) | 25 (26)
Headache (Nervous system disorders) | 18 (19) | 21 (24)
Subarachnoid haemorrhage (Nervous system disorders) | 16 (16) | 17 (17)
Haematoma (Vascular disorders) | 13 (13) | 1 (1)
Haemorrhagic infarction (Vascular disorders) | 20 (20) | 21 (21)
Hypotension (Vascular disorders) | 12 (12) | 17 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT03785678/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT03785678/SAP_001.pdf